CLINICAL TRIAL: NCT06611735
Title: The Effect of Retentive Rubber-Dam Clamps on Gingival Tissues During Restorative Treatment
Brief Title: Effect of Retentive Rubber-Dam Clamps
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2023.1296
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Gingival Health
Keywords: Direct restoration; gingival health; isolation; retention clamp; rubber-dam application

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retention clamp: Retention clamps applied to maxillary premolars during routine rubber dam isolation for performing anterior restorations.

SUMMARY:
This study aims to evaluate the effect of retention rubber dam clamps used on premolar teeth during rubber dam isolation on gingival health. The teeth to which retention clamps are applied were not undergo any restorative procedures. Retention clamps applied to maxillary premolars during routine rubber dam isolation for performing anterior restorations. Changes in periodontal tissues were evaluated; using plaque index, bleeding on probing, probing depth, keratinized gingiva, attached gingiva, relative gingival margin level and relative attachment levels after the procedure at different times (pre-restoration, after restoration, 1 week, 1 month, 3 month). The evaluation time was planned not to exceed 10 minutes, restorations are done by a single specialist in Marmara University Restorative Dentistry Department.

DETAILED DESCRIPTION:
In the present study, it is aimed to evaluate the effect of retention rubber dam clamps used on premolar teeth during rubber dam isolation on gingival health. The teeth to which retention clamps are applied were not undergo any restorative procedures. Retention clamps applied to maxillary premolars during routine rubber dam isolation for performing anterior restorations. The application time of the retention clamps were limited as maximum 2 hours. Before starting the treatment, patients signed information and consent forms. In the present study, direct composite restorations were planned under local anesthesia, and it was planned to evaluate the effects of retention clamps on periodontal tissues and patient comfort. After the isolation, direct composite restorations were performed.

- Data collection method Changes in periodontal tissues were evaluated; using plaque index, bleeding on probing, probing depth, keratinized gingiva, attached gingiva, relative gingival margin level, relative attachment level after the procedure at different times (pre-restoration, after restoration). It was evaluated immediately after, 1 week later, 1 month later, 3 months later. The evaluation time was planned not to exceed 10 minutes, restorations are done by a single specialist in Marmara University Restorative Dentistry Department.

Restorative materials used in the study; Nic Tone Thick (Dental Dam, Nic Tone, Romania) was used as a rubber-dam rubber cover for patients. In addition, sterile frames (Hu-Friedy Group, USA), forceps (Hu-Friedy Group, USA) and puncher (Hu-Friedy Group, USA) were used as rubber-dam instruments on patients. For gingival retention, Hu-Friedy Black Line 2X clamps (Hu-Friedy Group, USA) were used.

Clinical Index and Measurements Determination of Gingival Phenotype Evaluating the visibility of the silhouette of the periodontal probe inserted into the sulcus is a technique used to determine the phenotype. If the silhouette of the probe placed in the sulcus is visible, the gingiva is considered thin, and if it is not, the gingiva is considered thick.

Keratinized Gums The distance between the mucogingival junction and the gingival margin were measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.

Attached Gingiva The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.

Plaque Index For each tooth, plaque index measurements were made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.

Bleeding on Probing Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values were given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.

Probing Depth For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.

Relative Attachment Level Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement was made in 6 regions, mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces of each tooth.

Relative Gingival Margin Level Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual/palatinal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.

Evaluation of Restorations Restorations were evaluated according to FDI (Fédération Dentaire Internationale) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Have sufficient cognitive ability to understand the consent procedure
* Clinically healthy gingiva and periodontium
* Daily cigarette consumption of 10 or less
* No attachment loss, bleeding on probing, or plaque buildup
* Patients with cervical lesions, abrasion lesions and/or indications for diastema closure requiring restoration
* Patients with cervical lesions at or below the gingival level
* Patients with direct composite restoration indications concerning the anterior region.

Exclusion Criteria:

* Any disability (mental health conditions, mentally handicapped and physically handicapped)
* Systemic diseases or serious medical risks (Cardiovascular disorder, diabetes, hypertensive, epileptic)
* Compliance problem, inability to provide post-treatment hygiene
* Gingival hyperplasia or bleeding disorder
* Signs of attachment loss of periodontal disease
* Patients for whom rubber dam placement is contraindicated (patient with asthma diagnosis, mouth breathing, partially erupted tooth, overly malpositioned teeth and latex allergy).
* Signs of periapical pathology or pulpal posterior or anterior pathology
* Teeth which have mobility
* Teeth with extraction indication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who attended Marmara University Faculty of Dentistry Restorative Department, for the anterior restorations.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Measurement of plaque index before the treatment | Before the treatment
  For each tooth, plaque index measurements were made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.
Measurement of probing depth before the treatment | Before the treatment
  For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.
Measurement of bleeding on probing before the treatment | Before the treatment
  Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.
Measurement of keratinized gingiva before the treatment | Before the treatment
  The distance between the mucogingival junction and the gingival margin was measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.
Measurement of attached gingiva before the treatment | Before the treatment
  The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.
Measurement of relative gingival margin level before the treatment | Before the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 3 regions of each tooth: mesiobuccal, midbuccal, and distobuccal surfaces.
Measurement of relative attachment level before the treatment | Before the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 3 regions, mesiobuccal, midbuccal, distobuccal surfaces of each tooth.

SECONDARY OUTCOMES:
Measurement of probing depth immediately after the treatment | Immediately after the treatment
  For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.
Measurement of bleeding on probing immediately after the treatment | Immediately after the treatment
  Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.
Measurement of keratinized gingiva immediately after the treatment | Immediately after the treatment
  The distance between the mucogingival junction and the gingival margin was measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.
Measurement of attached gingiva immediately after the treatment | Immediately after the treatment
  The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.
Measurement of relative gingival attachment level immediately after the treatment | Immediately after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 3 regions, mesiobuccal, midbuccal, distobuccal surfaces of each tooth.
Measurement of relative gingival margin level immediately after the treatment | Immediately after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 3 regions of each tooth: mesiobuccal, midbuccal, and distobuccal surfaces.
Measurement of plaque index of 1 week control session | 1 week after the treatment
  For each tooth, plaque index measurements were made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.
Measurement of probing depth of 1 week control session | 1 week after the treatment
  For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.
Measurement of bleeding on probing of 1 week control session | 1 week after the treatment
  Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.
Measurement of keratinized gingiva of 1 week control session | 1 week after the treatment
  The distance between the mucogingival junction and the gingival margin was measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.
Measurement of attached gingiva of 1 week control session | 1 week after the treatment
  The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.
Measurement of relative gingival margin level of 1 week control session | 1 week after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 3 regions of each tooth: mesiobuccal, midbuccal, and distobuccal surfaces.
Measurement of relative attachment level of 1 week control session | 1 week after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 3 regions, mesiobuccal, midbuccal, distobuccal surfaces of each tooth.
Measurement of plaque index of 1 month control session | 1 month after the treatment
  For each tooth, plaque index measurements were made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.
Measurement of probing depth of 1 month control session | 1 month after the treatment
  For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.
Measurement of bleeding on probing of 1 month control session | 1 month after the treatment
  Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.
Measurement of keratinized gingiva of 1 month control session | 1 month after the treatment
  The distance between the mucogingival junction and the gingival margin was measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.
Measurement of attached gingiva of 1 month control session | 1 month after the treatment
  The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.
Measurement of relative gingival margin level of 1 month control session | 1 month after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 3 regions of each tooth: mesiobuccal, midbuccal, and distobuccal surfaces.
Measurement of relative attachment level of 1 month control session | 1 month after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 3 regions, mesiobuccal, midbuccal, distobuccal surfaces of each tooth.
Measurement of plaque index of 3 months control session | 3 months after the treatment
  For each tooth, plaque index measurements were made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.
Measurement of probing depth of 3 months control session | 3 months after the treatment
  For each of the initially selected teeth, probing depth measurements were made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.
Measurement of bleeding on probing of 3 months control session | 3 months after the treatment
  Bleeding on probing was examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.
Measurement of keratinized gingiva of 3 months control session | 3 months after the treatment
  The distance between the mucogingival junction and the gingival margin was measured as the width of the keratinized gingiva after the alveolar mucosa was pushed and curved coronally and with periodontal probe and the mucogingival junction was determined.
Measurement of attached gingiva of 3 months control session | 3 months after the treatment
  The distance between the mucogingival junction and the floor of gingival sulcus was measured as the width of the attached gingiva.
Measurement of relative gingival margin level of 3 months control session | 3 months after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the incisal guide and the gingival margin was measured and recorded. Relative gingival margin level measurement was made in a total of 3 regions of each tooth: mesiobuccal, midbuccal, and distobuccal surfaces.
Measurement of relative attachment level of 3 months control session | 3 months after the treatment
  Using the Chu's Gauge handpiece, it was placed on the incisal edge of the incisors, the incisal guide edge of the handpiece was taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge was measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 3 regions, mesiobuccal, midbuccal, distobuccal surfaces of each tooth.

CONTACTS AND LOCATIONS:
Overall Officials: EZGİ Tüter Bayraktar, Assistant Professor, Principal Investigator — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the article, data will be shared.
Supporting Information: Study Protocol, SAP